CLINICAL TRIAL: NCT05900908
Title: A Randomized Controlled Trial of Surgical Resection With GammaTile Therapy and Adjuvant Systemic Therapy Compared to Surgical Resection and Adjuvant Systemic Therapy at First Recurrence in Glioblastoma.
Brief Title: Post-operative Adjuvant Therapy w/wo GammaTile + Systemic Therapy
Acronym: PATHWAyS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study is being withdrawn in favor of a different study schema to be launched later this year.
Sponsor: GT Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GTM-104
Record Dates: First submitted 2023-05-25; First posted 2023-06-13 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Glioblastoma
Keywords: Brain; Tumor; Glioblastoma; Recurrent; Cancer; Metastases; GammaTile; Radiation; Cs-131
MeSH Terms: conditions — Glioblastoma; Neoplasms; Recurrence; Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- surgical tumor removal and GammaTile therapy followed by adjuvant systemic therapy (Experimental): surgical tumor removal and GammaTile therapy followed by adjuvant systemic therapy
  Interventions: Device: Gamma Tile-Surgically Targeted Radiation Therapy (STaRT)
- surgical tumor removal followed by adjuvant systemic therapy (Active Comparator): surgical tumor removal followed by adjuvant systemic therapy
  Interventions: Radiation: Stereotactic Radiation Therapy

INTERVENTIONS:
Device: Gamma Tile-Surgically Targeted Radiation Therapy (STaRT) — GammaTiles are a permanently implanted radiation device consisting of Cs-131 seeds positioned within a collagen tile
  Other Names: Carrier Tile Brachytherapy Therapy (CTBT)
  Arms: surgical tumor removal and GammaTile therapy followed by adjuvant systemic therapy
Radiation: Stereotactic Radiation Therapy — External Beam Radiation Therapy
  Arms: surgical tumor removal followed by adjuvant systemic therapy

SUMMARY:
To compare surgical tumor removal and GammaTile therapy followed by adjuvant systemic therapy (bevacizumab or lomustine) to surgical tumor removal followed by adjuvant systemic therapy (bevacizumab or lomustine) without GammaTile therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years old and above. Eligibility is restricted to this age group given that the battery of neurocognitive tests utilized in this protocol are not developed or validated for use in a younger population.
2. History of a histopathologically and molecularly confirmed glioblastoma, per Consortium to Inform Molecular and Practical Approaches to Central Nervous System Tumor Taxonomy (c-IMPACT-NOW) criteria ("diffuse astrocytic glioma, IDH-wildtype, with molecular features of glioblastoma, World Health Organization [WHO] grade IV"; this requires presence of amplification of EGFR, whole chromosome 7 gain AND whole chromosome 10 loss, or Telomerase reverse transcriptase (TERT) promoter mutation.
3. Patients for which bevacizumab or lomustine are reasonable systemic treatments following surgery.
4. Eligible patients must be experiencing a known or suspected first recurrence of a supratentorial GBM following prior first-line concurrent TMZ and RT (allowed hypofractionation of prior RT dose ≥ 40 Gray [Gy] of a planned 60 Gy dose) and at least one cycle of adjuvant TMZ. RT must have concluded >45 days prior to enrollment, and most recent adjuvant TMZ treatment(s) must have been concluded or terminated >10 days prior to enrollment. Prior adjuvant TMZ cycles up to 12, prior adjuvant tumor-treating fields (TTF), and prior External Beam Radiotherapy (EBRT) doses via proton or photon treatments up to 72 Gy equivalent are allowed. Note: This includes infratentorial recurrences of tumors that were supratentorial at diagnosis. Tumors the were infratentorial at diagnosis are excluded.
5. Eligible tumors are defined as the following:

   1. Supratentorial
   2. A bi-dimensionally measurable lesion of at least 10 mm, visible on two or more axial slices 5 mm apart.
   3. The pre-operative tumor (including enhanced and unenhanced tumor) planned for resection that is 60 mm2 or less in maximum cross section.
   4. Tumor that in the opinion of the enrolling neurosurgeon is amenable to attempted gross total resection (GTR). Prior diagnostic biopsy allowed.
   5. Anticipated GammaTile placement (i.e., closest aspect of post resection tumor bed that is anticipated to receive GammaTile placement) that is > 15mm from the optic chiasm or brainstem.
   6. Multifocal enhancing disease is allowed if it can be fully encompassed in one operative bed while meeting criterion a-e.
6. Ability to complete an MRI of the head with and without contrast, and a non-contrast CT.
7. All subjects fluent in English will complete neurocognitive evaluations. Patients not fluent in English are allowed on trial but will not take neurocognitive tests as comparative data is only available from tests in the English language.
8. Tumor O-6-methylguanine-deoxyribonucleic acid (DNA) methyltransferase (MGMT) methylation status must be available from any prior GBM tumor specimen; results of routinely used methods for MGMT methylation testing (e.g., mutagenically separated polymerase chain reaction [MSPCR] or quantitative polymerase chain reaction [PCR]) are acceptable and results can be from a local lab or central lab used by a prior study.
9. Suspicion of suspected tumor recurrence is on imaging and/or histologic grounds. If imaging, at a minimum a contrast-enhanced MRI scan ≤21 days prior to registration (at the time of randomization) should meet Response Assessment in Neuro-Oncology (RANO) criteria.
10. Concomitant systemic or local anti-cancer medications or treatments, other than those on this protocol, are prohibited in this study in the absence of progression.
11. Patients can be on a stable or decreasing dose of steroids for 1 week before the screening MRI. Utilization of the lowest useful dose and shortest useful course are encouraged.
12. Karnofsky Performance Scale (KPS) score of ≥ 70 documented within ± 21 days of signing consent.
13. Eastern Cooperative Oncology Group Performance Score (ECOG-PS) of <2 documented ≤ 21 days of signing consent.
14. Blood test results ≤ 21 days prior to surgery (can be re-run prior to surgery):

    1. Leukocytes ≥ 2,500/mm3
    2. Absolute neutrophil count ≥ 1,500/mm3
    3. Absolute lymphocyte count ≥ 800/mm3
    4. Platelets ≥ 75,000/mm3
    5. Hemoglobin ≥ 8 g/dL
    6. Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (however, patients with known Gilbert disease who have serum bilirubin level ≤ 3 x ULN may be enrolled)
    7. Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])

       * 2.5 x ULN
    8. Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x ULN
    9. Alkaline phosphatase ≤ 2.5 x ULN
    10. Creatinine clearance ≥ 50 mL/min/1.73 m2 by Cockcroft-Gault
15. Women of childbearing potential must have a negative serum or urine pregnancy test ≤7 days prior to randomization. Women must be willing to notify investigator immediately if they become pregnant at any time during the trial period. They must be willing to use a form of contraception to prevent pregnancy during treatment.
16. Willingness and ability to provide written informed consent or have their legally authorized representative provide consent and Health Insurance Portability and Accountability (HIPAA) authorization for them if they physically are unable to sign prior to performance of any study-related procedure.
17. Availability of prior radiotherapy treatment plan details in Digital Imaging and Communications in Medicine (DICOM) format is desired but not required for study participation.

Exclusion Criteria:

1. Any previous treatment for recurrent GBM.
2. Patients with suspected or confirmed radiation necrosis.
3. Known somatic tumor mutation in IDH1 or IDH2 gene. If not previously completed, sequencing of the IDH1 and IDH2 genes is not required to determine trial eligibility.
4. Known germline DNA repair defect (mismatch repair deficiency, POLE mutation, e.g.). If not previously completed, germline sequencing is not required to determine trial eligibility.
5. Patients not appropriate for treatment with bevacizumab or lomustine, in the opinion of the investigator or medical team.
6. Patients for whom any additional treatment is planned in the absence of recurrent or progressive disease.
7. Leptomeningeal disease not expected to be encompassed by the surgical resection.
8. History of treatment with carmustine implants (Gliadel)
9. Previous or concurrent bevacizumab therapy for treatment of tumor. Use of bevacizumab is allowed for reducing edema. Must be off of bevacizumab for at least 28 days prior to surgery.
10. If bevacizumab is pre-planned for adjuvant systemic treatment, the following contraindications to the use of bevacizumab, must be absent. (Note: If any of these contraindications exist, the use of lomustine must be considered as the systemic agent. If both bevacizumab and lomustine are inappropriate in the treating physician's opinion, the patient must be excluded).
11. Clinically Significant Cardiovascular Disease Defined as follows: Inadequately controlled hypertension (i.e., systolic blood pressure (SBP) > 160 mm Hg and/or diastolic blood pressure (DBP) > 90 mm Hg despite antihypertensive therapy).

    1. History of cerebrovascular accident (CVA) ≤ 180 days.
    2. Myocardial infarction or unstable angina ≤ 180 days.
    3. Pulmonary embolism ≤180 days
    4. Evidence or history of bleeding diathesis (greater than normal risk of bleeding, i.e., Hereditary Hemorrhagic Telangiectasia Type I or HHT-1) or coagulopathy in the absence of therapeutic anti-coagulation or any hemorrhage/bleeding event > Grade 3

       * 28 days prior to registration. Note: Patients with full-dose anticoagulants are eligible provided the patient has been on a stable dose for ≥14 days.
12. Active wound, a serious or non-healing wound, an active ulcer or untreated bone fracture.
13. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess ≤ 180 days prior to consenting.
14. Previous or current treatment with an investigational or FDA approved systemic therapy for glioblastoma other than external beam radiation (proton or photon), temozolomide (Temodar®), or tumor treatment fields (Optune®) (e.g., other forms of systemic therapy, targeted therapeutics, immunotherapy).
15. Sensitivity to bovine (cow) derived materials including collagen products.
16. Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen are excluded from this trial.
17. Severe infections ≤ 21 days prior to signing consent including, but not limited to, hospitalization for complications of infection, bacteremia, viral infections (COVID-19 [Corona Virus Disease 2019], Hepatitis B or C, Human Immunodeficiency Virus [HIV]) or severe pneumonia.
18. Major surgical procedure ≤21 days prior to protocol surgery or anticipation of need for a major surgical procedure during the course of study treatment.
19. Uncontrolled intercurrent illness including, but not limited to, uncontrolled hypertension (systolic blood pressure >140 mm Hg or diastolic blood pressure >90 mm Hg) despite optimal medical management; myocardial infarction less than 6 months before the planned surgery date; arterial thrombotic or embolic events, such as cerebrovascular accident (including transient ischemic attacks) or pulmonary embolism 180 days before the planned surgery date, or psychiatric illness/social situations that would impair understanding or limit compliance with study requirements, including ability to complete neurocognitive assessments and quality of life questionnaires, and returning for follow-up care
20. Any concomitant therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
21. Women who are pregnant or nursing are excluded from this study.
22. Patients who experienced a toxicity of grade ≥ 3 (CTCAE v5) from prior GBM treatment, unless they have sufficiently recovered as evidenced by a drop to grade ≤2 or have full resolution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Median Overall Survival (OS) from the time of surgery up to 2 years post surgery. | up to 2 years
  Analysis of primary outcome measure will include the intent to treat population.

SECONDARY OUTCOMES:
Overall Survival | up to 2 years
  A measure of median overall survival for the per protocol population
Progression free survival (PFS) | up to 2 years
  A measure of time from surgery to any failure, local or distant.
Change in Quality of Life (QOL) | up to 1.5 years
  Functional Assessment of Cancer Therapy-Brain (FACT-Br)
Assessment of Neurocognitive Function | up to 1.5 years
  Hopkins Verbal Learning Test-Revised [HVLT-R]
Functional Status-Karnofsky Performance Scale (KPS) | up to 2 years
  An assessment of functional impairment. Score 0 to 100, with 100 being no impairment of performance
Proportion of subjects with evidence of radiation necrosis (RN) | up to 2 years
  A measure of patients who experience radiation necrosis post-surgery.
Proportion of subjects with evidence of surgical site wound infection | Up to 1.5 months
  A measure of patients who experience surgical site wound infection
Proportion of subjects with evidence of a surgical site dural closure-related cerebral spinal fluid (CSF) leak | Up to 1.5 months
  A measure of patients who experience surgical site dural closure-related cerebral spinal fluid (CSF) leak
Post-surgery length of hospital stay of study subjects | Up to 1.5 months
  A measure in days of the length of hospital stay post surgery.
Rate of re-admission | Up to 1 month
  A measure of patients re-admitted to the hospital +/- 30 days post surgery.

IPD SHARING:
Plan to Share IPD: No